CLINICAL TRIAL: NCT04578977
Title: Evaluation of Surgical Treatment of Terrible Triade Injury of the Elbow Joint
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, abdalraouf mahmoud ghozaly, Evaluation of Surgical Treatment of Terrible Triade Injury of the Elbow joint, Assiut University
Other Study IDs: Treatment of Terrible Triade
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Treatment of Terrible Triade Injury of the Elbow Joint

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Functional assessment of surgical treatment of terrible triade injury of the elbow — Functional assessment of surgical treatment of terrible triade injury of the elbow

SUMMARY:
) Terrible triad injury of the elbow is a complex injury that is classically defined as elbow dislocation along with fractures of the coronoid process of the ulna and the radial head. The injury is usually associated with typical soft-tissue disruptions (with common involvement of the lateral collateral ligament complex, elbow joint capsule, as well as the common extensor and flexor-pronator tendons)(2).

Complications of terrible triad injuries include redislocation, residual instability, elbow stiffness, heterotopic ossification, fracture malunion or nonunion, elbow arthrosis, olecranon bursitis, ulnar or radial nerve palsy (due to the surgical approach or placement of hardware), and hardware related complications(2) .

Management of trrible triade is conservative or surgical treatment ,in this study we will use surgical treatment and make evaluation of it.

DETAILED DESCRIPTION:
The elbow is the second most commonly dislocated joint in adults and up to 20% of dislocations are associated with a fracture. (1) Terrible triad injury of the elbow is a complex injury that is classically defined as elbow dislocation along with fractures of the coronoid process of the ulna and the radial head. The injury is usually associated with typical soft-tissue disruptions (with common involvement of the lateral collateral ligament complex, elbow joint capsule, as well as the common extensor and flexor-pronator tendons) Complications of terrible triad injuries include redislocation, residual instability, elbow stiffness, heterotopic ossification, fracture malunion or nonunion, elbow arthrosis, olecranon bursitis, ulnar or radial nerve palsy (due to the surgical approach or placement of hardware), and hardware related complications.

Management of trrible triade is conservative or surgical treatment ,in this study we will use surgical treatment and make evaluation of it.

Surgical treatment involves radial head repair or replacement ,medial and lateral collateral ligament repair and coronoid fracture fixation.

aim of research isFunctional assessment of surgical treatment of terrible triade injury of the elbow according to Mayo elbow performance score, According to the system of Mayo, scores of 90-100 are classified as excellent, 75-89 as good, 60-74 as fair, and 0-59 as poor

ELIGIBILITY:
Inclusion Criteria:

* 1.skeletally mature patients (over 17 years old) including both sexes. 2.Acute fractures within 3 weeks of injury. 3.Isolated & closed fractures . 4.polytrauma trauma patients with no other injuries in the same limb.

Exclusion Criteria:

* 1. pathological fracture of proximal radius and ulna. 2. deteriorateed general health. 3. previous history of dysfunction with the affected elbow.

Min Age: 17 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: clinical case series study .
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-10-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Surgical Treatment of Terrible Triade Injury of the Elbow joint. | 2 years
  Functional assessment of surgical treatment of terrible triade injury of the elbow according to Mayo elbow performance score

CONTACTS AND LOCATIONS:
Overall Officials: Abdalraouf Mahmoud Ghozaly, resident doctor, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Kani KK, Chew FS. Terrible triad injuries of the elbow. Emerg Radiol. 2019 Jun;26(3):341-347. doi: 10.1007/s10140-019-01676-1. Epub 2019 Jan 28. PMID 30690677
- [Result] Jones ADR, Jordan RW. Complex Elbow Dislocations and the "Terrible Triad" Injury. Open Orthop J. 2017 Nov 30;11:1394-1404. doi: 10.2174/1874325001711011394. eCollection 2017. PMID 29290879